CLINICAL TRIAL: NCT04807075
Title: A Wearable, Battery-free Screening System for SARS-CoV-2, the Virus Causing COVID-19 Infection
Status: Terminated | Type: Observational
Why Stopped: Failure to recruit
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0027-21-EP
Record Dates: First submitted 2021-03-17; First posted 2021-03-19 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The corona virus disease (COVID) pandemic has highlighted the importance of rapid, readily available screeners and diagnostics to identify infected individuals. Recent studies have demonstrated that portable electronic nose sensing devices can detect volatile organic compounds (VOCs). These compounds are end products of human metabolism or of enteric bacteria and are excreted through the skin or exhaled breath. Importantly, the sensing devices can be adapted into a wearable device providing continuous monitoring. Our goal is to develop a battery-free, electronic nose sensor to serve as a screener and detect VOC patterns associated to patients with symptomatic and asymptomatic COVID-19 without being invasive. To test the screening ability, devices will be worn by COVID-19 positive and negative patients hospitalized at Nebraska Medicine.

DETAILED DESCRIPTION:
Purpose. This study will assess the feasibility of using an electronic nose to detect signals indicating infection with severe acute respiratory distress syndrome corona virus-2 (SARS-CoV-2). Five different prototypes of electronic nose will be used that would be deployed differently: 1) a patch, 2) clipped to a garment neckline, 3) clipped to a garment waistline, 4) resting on a bedside table, and 5) integrated into a facemask. Data will be collected over a three day period to determine the quality of the smell-print signals collected by the different deployment regimes. Eligibility. Subjects admitted to University of Nebraska Medical Center (UNMC) with definite or suspected SARS-CoV-2 infection will be eligible. Subjects must have access to a smart phone and be well enough to engage in the active data collection. The goal is to enroll 30 SARS-CoV-2 infected and 30 uninfected individuals. Eligibility of controls will be extended to patients admitted to UNMC with other respiratory problems including chronic obstructive pulmonary disease (COPD) exacerbation, pneumonia and congestive heart failure if needed. Adults (19 years and older) are eligible. Subjects with allergic reactions to components of the devices will be excluded. Interventions and evaluations. Informed consent will be obtained remotely following which an app will be downloaded to their phone. A kit will be delivered to the patients room containing the five devices. The app will support: instruction on use of the devices, reminders to collect data every 2 hours between 08:00 and 20:00, and access to study personnel for support as needed. The app will transmit smell prints from the 5 devices to a secure cloud-based database. The study coordinator will oversee subject education and deployment of the devices by phone/facetime. Subjects will be instructed on use of the devices, which they will self-deploy in positions that do not interfere with any medical equipment. The patch, clip-ons and bedside sensor will be worn continuously from 08:00 to 20:00. The mask will be placed for 5 minutes before each data collection, which will be timed by the phone app. The mask can then be removed until the next data collection. Smell-print data will be collected for three days. Following this, the devices will be replaced into the kit box and collected by the nursing staff. Clinical data will be collected from the electronic health record. Follow up. Following completion of the study, subjects will be asked to complete a brief questionnaire on the experience and asked about their willingness to be contacted for further interviews.

ELIGIBILITY:
Inclusion Criteria:

°Admission for definite or suspected SARS-CoV-2 infection with mild to moderate symptoms and clinical features.

If insufficient numbers of suspected cases who test negative, individuals admitted with other respiratory problems: COPD exacerbation, viral pneumonia, congestive heart failure who test negative for SARS-CoV-2 will be eligible as controls.

* Able to give informed consent.
* Access to a smartphone capable of downloading the study app and of collecting and transmitting study data.
* Ability to comply with study procedures.
* Ability to self-deploy the study devices and collect study data.

Exclusion Criteria:

* Inability to give informed consent.
* Allergic history to components of study devices,
* Inability to participate in study procedures.
* Severe disease or admission to a critical care unit.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (age >18) subjects admitted to the hospital for possible COVID-19.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2021-04-04 (Actual); Primary Completion 2022-06-07 (Actual); Study Completion 2022-06-07 (Actual)

PRIMARY OUTCOMES:
nose smell-print | at enrollment
  nose smell-print. This is recorded as a set of impedances, one from each sensor filament. This results in an 8-dimensional vector that will be recorded for each subject. The vectors will then be related to diagnostic category (SARS-CoV-2 positive vs. negative). This will be determined separately for each of the sensor devices.

SECONDARY OUTCOMES:
stability of smell print | three days
  8-dimensional smell prints will be recorded at approximately 2 hour intervals for waking hours over three days.

CONTACTS AND LOCATIONS:
Overall Officials: Chad L Vokoun, MD, Principal Investigator — UNMC
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No